CLINICAL TRIAL: NCT06812143
Title: Optimizing Strength Training in Older Adults
Acronym: LOAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queens College, The City University of New York (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anoop T Balachandran, Assistant Professor, Queens College, The City University of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R15AG085170 (NIH); 1R15AG085170-01 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Aging
Keywords: Strength training; Older adults; physical function
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light Load, High Repetition (LLHR) (Experimental): The LLHR group will perform a full-body routine with lighter weights, performing 16-20 repetitions per set, close to failure.
  Interventions: Behavioral: Strength training
- Strength Training (ST) (Active Comparator): The ST group will perform a full-body routine with higher weights, performing 8-12 repetitions per set, close to failure.
  Interventions: Behavioral: Strength training

INTERVENTIONS:
Behavioral: Strength training — This intervention involves strength training with lighter loads and higher repetitions.
  Other Names: Resistance training; Weight training
  Arms: Light Load, High Repetition (LLHR)
Behavioral: Strength training — This intervention involves conventional strength training with higher loads and moderate repetitions.
  Other Names: Resistance trainig; Weight training
  Arms: Strength Training (ST)

SUMMARY:
The objective of the current study is to determine whether lifting lighter loads close to failure improves strength training adaptations and function in older adults. The main questions it aims to answer are:

1. The effect of light loads on physical function
2. The effect of light loads on muscle mass, power, and strength

Researchers will compare a light-load, high-repetition program to a standard strength training program. Participants will perform supervised strength training twice per week for 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 65 years and above
* Inactive lifestyle (< 150 min per week of moderate intensity physical activity) and not regularly participating in a structured strength training program
* Planning to reside in the area for the duration of the study

Exclusion Criteria:

* Severe cardiac disease, including Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Lung disease requiring either oral or injected steroids, or the use of supplemental oxygen
* Short, portable mental status questionnaire with 3 or more errors
* Severe arthritis (either osteoarthritis or rheumatoid arthritis)
* Cancer requiring treatment in the past 1 year (melanomas excluded)
* Development of chest pain or severe shortness of breath during the 6 min self-paced walk test
* Parkinson's disease or other serious neurological disorders
* Renal disease requiring dialysis
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Current consumption of more than 14 alcoholic drinks per week
* Severe lower back or shoulder pain that may worsen with weightlifting exercises
* Undergoing physical therapy involving the lower extremities
* Living in nursing homes, assisted living facilities or other similar institutions
* Currently enrolled in another randomized trial involving a pharmaceutical or lifestyle intervention
* Weight change (intentional or not) over the last 6 months of > 5% of body weight, or plan to lose or gain weight during the study
* Any other cardiovascular, pulmonary, orthopedic, neurologic, or other conditions that would preclude participation and successful completion of the protocol

Temporary Exclusion Criteria

A person meeting any of the following temporary exclusion criteria at the time of screening will not be enrolled but may be re-screened later.

* Severe hypertension, e.g., SBP > 200 mm Hg, DBP > 110 mm Hg
* Major surgery or fracture or hip/knee replacement within the last 6 months
* Hospitalization within the last 6 months (excluding ER visits)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | Baseline and week 21
  Change in the total distance walked in 6 minutes. The 6-minute walk test is an objective, well-validated, and clinically meaningful measure of physical function in older adults.

SECONDARY OUTCOMES:
Lower body maximal muscle strength | Baseline and week 21.
  Change in lower body maximum muscle strength will be assessed using a one-repetition maximum (1RM) test on a leg press machine.
Lower body muscle power | Baseline and week 21
  Lower body muscle peak power (W) will be assessed using a pneumatic leg press machine.
Lean body mass (LBM) | Baseline and week 21
  Change in total lean body mass (kg) will be assessed using a dual-energy X-ray absorptiometry (DXA) scan
Self-reported physical function | Baseline and week 21
  Self-reported physical function will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) physical function questionnaire. PROMIS measures are scored on the T-score metric. High scores mean more of the concept being measured.
Get-up & go test | Baseline and week 21
  Change in the time (in seconds) taken to complete the get up and go test. The get up & go test will be used to assess lower body dynamic balance and fall risk
30-second chair stand test | Baseline and week 21
  Change in the number of repetitions completed during the 30-Second chair stand test. This test assesses lower body functional strength and power.
Number of participants with adverse events | From enrollment to the end of 20-week intervention period
  Number of participants experiencing adverse events that are possibly or definitely related to the intervention,
Physical activity enjoyment scale (PACES) | Week 21
  Participants will complete the 18-item Physical activity enjoyment scale (PACES) to assess their level of physical activity enjoyment. Scores range from 18 to 126 and higher scores indicate greater enjoyment.
Exercise self-efficacy questionnaire | Week 21
  Participants will complete the exercise self-efficacy scale to assess their belief in their ability to continue strength training twice per week at the prescribed intensity in the future. Scores range from 0 to 100 and higher scores indicate greater self-efficacy.
Exercise session attendance | From enrollment to the end of 20-week intervention period
  The total number of supervised exercise sessions attended by participants over the 20-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise & Aging Lab, Queens College, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] T Balachandran A, Wang Y, Szabo F, Watts-Battey C, Schoenfeld BJ, Zenko Z, Quiles N. Comparison of traditional vs. lighter load strength training on fat-free mass, strength, power and affective responses in middle and older-aged adults: A pilot randomized trial. Exp Gerontol. 2023 Jul;178:112219. doi: 10.1016/j.exger.2023.112219. Epub 2023 May 30. PMID 37236327